CLINICAL TRIAL: NCT02702271
Title: Protection Against Embolism for Non-valvular AF Subjects: Investigational Device Evaluation of the WATCHMAN FLX™ LAA Closure Technology
Brief Title: Investigational Device Evaluation of the WATCHMAN FLX™ LAA Closure Technology
Acronym: PINNACLE FLX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 91081206
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A total of 400 main cohort subjects and 58 roll-in subjects were enrolled at 29 investigational centers in the United States.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- WATCHMAN FLX - M (Experimental): WATCHMAN FLX Main Cohort
  Interventions: Device: WATCHMAN FLX
- WATCHMAN FLX - R (Experimental): WATCHMAN FLX Roll-In Cohort
  Interventions: Device: WATCHMAN FLX

INTERVENTIONS:
Device: WATCHMAN FLX — Left atrial appendage closure with WATCHMAN FLX

SUMMARY:
The study is a prospective, non-randomized, multi-center investigation to establish the safety and effectiveness of the WATCHMAN FLX™ Left Atrial Appendage Closure Device for subjects with non-valvular atrial fibrillation who are eligible for long-term anti-coagulation therapy to reduce the risk of stroke but who have a rationale to seek a non-pharmacologic alternative.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years of age or older.
2. The subject has documented paroxysmal, persistent, permanent or long-term/longstanding persistent non-valvular atrial fibrillation (i.e., the subject has not been diagnosed with rheumatic mitral valvular heart disease).
3. The subject is eligible for the defined protocol pharmacologic regimen of anticoagulation and antiplatelet therapy following WATCHMAN FLX Device implant.
4. The subject is eligible to come off of anticoagulation therapy if the LAA is sealed (i.e., the subject has no other conditions that would require long-term anticoagulation therapy suggested by current standard medical practice).
5. The subject has a calculated CHA2DS2-VASc score of 2 or greater for males or 3 or greater for females.
6. The subject is able to understand and willing to provide written informed consent to participate in the trial.
7. The subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

1. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility, regardless of type of co-enrollment being proposed.
2. The subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction, for example due to an underlying hypercoaguable state (i.e., even if the device is implanted, the subjects would not be eligible to discontinue anticoagulation due to other medical conditions requiring chronic anticoagulation therapy).
3. The subject is contraindicated for short-term anticoagulant therapy with DOAC post-implant.
4. The subject is contraindicated to aspirin and/or clopidogrel.
5. The subject is indicated for clopidogrel therapy or has taken clopidogrel within 7 days prior to the WATCHMAN FLX Device implant.
6. The subject had or is planning to have any cardiac or non-cardiac invasive or surgical procedure within 30 days prior to or 60 days after the WATCHMAN FLX Device implant (including, but not limited to: cardioversion, coronary angiogram with or without percutaneous coronary intervention (PCI), cardiac ablation, cataract surgery, endoscopy, etc.).
7. The subject had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within the 90 days prior to enrollment.
8. The subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 90 days prior to enrollment.
9. The subject has a history of atrial septal repair or has an ASD/PFO device.
10. The subject has an implanted mechanical valve prosthesis in any position.
11. The subject currently has New York Heart Association Class IV Congestive Heart Failure at the time of enrollment.
12. The subject is of childbearing potential and is, or plans to become pregnant during the time of the study (method of assessment upon study physician's discretion).
13. The subject has a documented life expectancy of less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shephal Doshi, MD, Principal Investigator — St. John's Health Center; Saibal Kar, MD, Principal Investigator — Los Robles Regional Medical Center
Locations (29):
- United States (29):
  - Grandview Medical Center, Birmingham, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Nair Research, LLC, Jonesboro, Arkansas
  - Scripps Green, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sharpe Chula Vista Medical Center, San Diego, California
  - St. John's Hospital / Pacific Heart, Santa Monica, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Cardiology Associates of N. Mississippi, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - New York University Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - York Hospital, York, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - PeaceHealth Southwest Medical, Vancouver, Washington

REFERENCES:
- [Derived] Kar S, Doshi SK, Sadhu A, Horton R, Osorio J, Ellis C, Stone J Jr, Shah M, Dukkipati SR, Adler S, Nair DG, Kim J, Wazni O, Price MJ, Asch FM, Holmes DR Jr, Shipley RD, Gordon NT, Allocco DJ, Reddy VY; PINNACLE FLX Investigators. Primary Outcome Evaluation of a Next-Generation Left Atrial Appendage Closure Device: Results From the PINNACLE FLX Trial. Circulation. 2021 May 4;143(18):1754-1762. doi: 10.1161/CIRCULATIONAHA.120.050117. Epub 2021 Apr 6. PMID 33820423

RESULTS

PARTICIPANT FLOW:
Groups:
- WATCHMAN FLX - M: Main Cohort
  WATCHMAN FLX: Left atrial appendage closure with WATCHMAN FLX
- WATCHMAN FLX - R: Roll-In Cohort
  WATCHMAN FLX: Left atrial appendage closure with WATCHMAN FLX
Period: Overall Study
Arm/Group | WATCHMAN FLX - M | WATCHMAN FLX - R
Started | 400 | 58
Completed | 337 | 49
Not Completed | 63 | 9
Not completed — Death | 36 | 7
Not completed — Lost to Follow-up | 12 | 0
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Unsuccessful Implant Attempt | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WATCHMAN FLX - M | WATCHMAN FLX - R | Total
Number analyzed (Participants) | 400 | 58 | 458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 7 | 62
  >=65 years | 345 | 51 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (8.6) | 75.2 (8.5) | 74.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 24 | 166
  Male | 258 | 34 | 292
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 10
  Not Hispanic or Latino | 390 | 58 | 448
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 2 | 20
  White | 358 | 51 | 409
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 5 | 26
Region of Enrollment [Number; unit: participants]
  United States | 400 | 58 | 458

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Safety Event
Description: The occurrence of one of the following events : all-cause death, ischemic stroke, systemic embolism, or device- or procedure-related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair. Percutaneous catheter drainage of pericardial effusions, snaring of an embolized device, thrombin injection to treat femoral pseudoaneurysm and nonsurgical treatments of access site complications are captured as adverse events (AEs), and are excluded from this endpoint.
Time Frame: events occurring between the time of implant and 7 days post procedure or by discharge, up to 30 days, whichever is later
Measure: Count of Participants; unit: Participants
Arm/Group | WATCHMAN FLX - M | WATCHMAN FLX - R
Number analyzed (Participants) | 400 | 58
Participants | 2 | 0

2. Primary Outcome: Number of Participants With Effective LAA Closure
Description: The rate of effective LAA closure, defined as any peri-device flow with jet size ≤ 5mm per core laboratory-assessed TEE at 12 months.
Time Frame: 12-months
Population: The Primary Effectiveness Endpoint is the rate of effective LAA closure at 12 months (defined as any peri-device flow with jet size ≤ 5mm per core laboratory-assessed TEE). The overall number of participants analyzed (342 in main and 52 in roll-in cohort) are the number of participants who had evaluable 12 month core lab f/u data from the total number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | WATCHMAN FLX - M | WATCHMAN FLX - R
Number analyzed (Participants) | 342 | 52
Participants | 342 | 52

ADVERSE EVENTS:
Time Frame: Adverse events that occur through 24 months post procedure.
Arm/Group | WATCHMAN FLX - M | WATCHMAN FLX - R
All-Cause Mortality (participants affected / at risk) | 36/400 | 7/58
Serious Adverse Events (participants affected / at risk) | 157/400 | 25/58
Other Adverse Events (participants affected / at risk) | 96/400 | 15/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN FLX - M (N=400) | WATCHMAN FLX - R (N=58)
Anaemia (Blood and lymphatic system disorders) | 11 (13) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 36 (38) | 3 (4)
Atrial flutter (Cardiac disorders) | 7 (8) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (6) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 7 (7) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 15 (22) | 6 (6)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 4 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (6) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 8 (9) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 15 (16) | 8 (9)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0)
Device related thrombosis (General disorders) | 6 (6) | 2 (2)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Multimorbidity (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (2)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Nocardiosis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 1 (3) | 0 (0)
Pneumonia (Infections and infestations) | 18 (19) | 4 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 10 (11) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subacute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 2 (2) | 0 (0)
Influenza B virus test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (2)
Device leakage (Product Issues) | 10 (12) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (6) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN FLX - M (N=400) | WATCHMAN FLX - R (N=58)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect acquired (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac steatosis (Cardiac disorders) | 1 (1) | 0 (0)
Chordae tendinae rupture (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 10 (10) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital oesophageal anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac complication associated with device (General disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 2 (2)
Catheter site haematoma (General disorders) | 3 (3) | 0 (0)
Catheter site haemorrhage (General disorders) | 7 (7) | 0 (0)
Catheter site vesicles (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cardiac septal defect residual shunt (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 14 (16) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (8) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Haematoma (Vascular disorders) | 5 (6) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT02702271/Prot_SAP_000.pdf